CLINICAL TRIAL: NCT01905605
Title: Phosphatidylcholine Supplementation in Infants With Diminished Sensory Gating
Brief Title: Phosphatidylcholine Supplementation in Infants
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding not secured. IRB approval has been withdrawn as of January 2017.
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13-2182
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Schizophrenia; Diminished P50 Sensory Gating
MeSH Terms: conditions — Schizophrenia | interventions — Phosphatidylcholines; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- phosphatidylcholine supplementation (Experimental): Phosphatidylcholine supplementation to be administered BID for 8 weeks
  Interventions: Drug: phosphatidylcholine supplementation
- placebo supplementation (Placebo Comparator): Placebo to be administered BID for 8 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: phosphatidylcholine supplementation — phosphatidylcholine concentrate 700 mg twice per day
  Other Names: Phosphatidylcholine, phosphatidylcholine concentrate
  Arms: phosphatidylcholine supplementation
Drug: placebo — placebo manufactured look like phosphatidylcholine concentrate dosed at 1.2 ml twice per day
  Other Names: Corn Oil
  Arms: placebo supplementation

SUMMARY:
Sensory gating is defined as the automatic process of inhibiting brain response to repeated auditory sounds. Infants who brains respond similarly to two identical sounds presented about 1/2 second apart are more likely to have later problems with attention than infants who suppress response to the second sound. This study will examine whether providing a nutritional supplement, phosphatidylcholine, for two months in infancy will result in an increased likelihood of developing more robust sensory gating.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infant has an age (adjusted for gestational age at birth) of 1-7 weeks
* Diminished P50 sensory gating (ratio greater than or equal to 0.50)

Exclusion Criteria:

* No maternal reported tobacco use for greater than 1 year and no current tobacco use (as measured by urine cotinine levels)
* Trimethylaminuria, renal disease, liver disease, known chromosomal abnormality, chronic neurological disorder, premature birth, prenatal exposure to exogenous steroid use

Ages: 1 Week to 7 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-09 (Estimated); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Ratio of P50 auditory sensory gating | 8 weeks post initiation of treatment
  In an auditory evoked potential paradigm while in active sleep (the infant equivalent of rapid eye movement sleep) with two identical sounds presented 500 ms apart, the ratio of the amplitude of the P50 response to the second sound divided by the amplitude of the P50 response to the first sound.

SECONDARY OUTCOMES:
Incidence of adverse events | 4 weeks and 8 weeks after initiation of intervention
  Percentage of infants with adverse events

OTHER OUTCOMES:
Percentage of planned dietary supplement | 8 weeks
  Percentage of planned dietary supplement given to the infant
Change in serum choline, betaine, and dimethylglycine levels | Randomization and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert Freedman, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States